CLINICAL TRIAL: NCT02446964
Title: Phase I Study of Escalating Doses of Total Marrow and Lymphoid Irradiation (TMLI) During Conditioning for HLA-Haploidentical Hematopoietic Cell Transplantation With Post-Transplant Cyclophosphamide in Patients With Myelodysplasia or Acute Leukemia
Brief Title: Total Marrow and Lymphoid Irradiation and Chemotherapy Before Donor Transplant in Treating Patients With Myelodysplastic Syndrome or Acute Leukemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14106; NCI-2015-00788 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 114382; 14106 (Other: City of Hope Medical Center)
Record Dates: First submitted 2015-05-14; First posted 2015-05-18 (Estimated); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: Adult Acute Lymphoblastic Leukemia in Complete Remission; Acute Myeloid Leukemia in Remission; Previously Treated Myelodysplastic Syndrome; Recurrent Adult Acute Lymphoblastic Leukemia; Recurrent Adult Acute Myeloid Leukemia; Recurrent Childhood Acute Lymphoblastic Leukemia; Recurrent Childhood Acute Myeloid Leukemia; Childhood Acute Lymphoblastic Leukemia in Complete Remission
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute | interventions — Bone Marrow Transplantation; Cyclophosphamide; fludarabine phosphate; Mycophenolic Acid; Peripheral Blood Stem Cell Transplantation; Tacrolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (TMLI, chemotherapy, transplant, GVHD prophylaxis) (Experimental): CONDITIONING: Patients undergo TMLI BID on days -7 to -4 or -3 (depending on the dose level). Patients also receive fludarabine phosphate IV on days -7 to -3 and cyclophosphamide IV on days -7, -6, 3, and 4.
  TRANSPLANT: Patients undergo bone marrow or peripheral blood stem cell transplant on day 0.
  GHVD PROPHYLAXIS: Patients receive tacrolimus* IV QD or PO BID on days 5-180. Patients also receive mycophenolate mofetil PO TID or IV on days 5-35. Treatment with tacrolimus and mycophenolate mofetil may continue in the presence of active GVHD.
  *NOTE: Patients intolerant of tacrolimus may receive cyclosporine.
  Interventions: Procedure: Bone Marrow Transplantation; Drug: Cyclophosphamide; Drug: Fludarabine Phosphate; Other: Laboratory Biomarker Analysis; Drug: Mycophenolate Mofetil; Procedure: Peripheral Blood Stem Cell Transplantation; Drug: Tacrolimus; Radiation: Total Marrow Irradiation

INTERVENTIONS:
Procedure: Bone Marrow Transplantation — Undergo bone marrow transplant
  Other Names: BMT; Bone Marrow Grafting; Bone Marrow Transplant; Marrow Transplantation
Drug: Cyclophosphamide — Given IV
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR- 138719
Drug: Fludarabine Phosphate — Given IV
  Other Names: 2-F-ara-AMP; 9H-Purin-6-amine, 2-fluoro-9-(5-O-phosphono-.beta.-D-arabinofuranosyl)-; Beneflur; Fludara; Oforta; SH T 586
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Mycophenolate Mofetil — Given PO or IV
  Other Names: Cellcept; MMF
Procedure: Peripheral Blood Stem Cell Transplantation — Undergo peripheral blood stem cell transplant
  Other Names: PBPC transplantation; Peripheral Blood Progenitor Cell Transplantation; Peripheral Stem Cell Support; Peripheral Stem Cell Transplantation
Drug: Tacrolimus — Given IV and PO
  Other Names: FK 506; Fujimycin; Prograf; Protopic
Radiation: Total Marrow Irradiation — Undergo TMLI

SUMMARY:
This phase I trial studies the side effects and best dose of total bone marrow and lymphoid irradiation when given together with chemotherapy before donor stem cell transplant in treating patients with myelodysplastic syndrome or acute leukemia. Total marrow and lymphoid irradiation is a type of radiation therapy that targets bone marrow and blood, where the cancer is, instead of applying radiation to the whole body. Stem cell transplants use high doses of chemotherapy and radiation therapy, such as total marrow and lymphoid irradiation, to kill cancer cells, but these treatments kill normal cells as well. After chemotherapy, healthy cells from a donor are given to the patient to help the patient grow new blood cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To establish safety and determine the maximum tolerated dose of total marrow and lymphoid irradiation when given in combination with fludarabine (fludarabine phosphate) and pre-post-transplant cyclophosphamide, as conditioning for haploidentical hematopoietic cell transplantation (HCT) in patients with high-risk acute lymphocytic or myelogenous leukemia or intermediate/high-risk myelodysplastic syndrome.

II. To evaluate the safety of the regimen at each dose level by assessing adverse events: type, frequency, severity, attribution, time course, duration.

III. To evaluate the safety of the regimen at each dose level by assessing complications: including acute/chronic graft-versus-host disease (GvHD), infection and delayed engraftment.

SECONDARY OBJECTIVES:

I. To estimate overall survival (OS), progression-free survival (PFS), cumulative incidence (CI) of relapse/progression, and non-relapse mortality (NRM) at +100 Days, 1 year and 2 years.

II. To characterize minimal residual disease from bone marrow aspirates on Days +30, +100, +180 post-transplant and describe in relation to total marrow and lymphoid irradiation (TMLI) dose level and patient disease status.

III. To describe the kinetics of immune cell recovery in the first year post-transplantation.

OUTLINE: This is a dose-escalation study of TMLI.

CONDITIONING: Patients undergo TMLI twice daily (BID) on days -7 to -4 or -3 (depending on the dose level). Patients also receive fludarabine phosphate intravenously (IV) on days -7 to -3 and cyclophosphamide IV on days -7, -6, 3, and 4.

TRANSPLANT: Patients undergo bone marrow or peripheral blood stem cell transplant on day 0.

GHVD PROPHYLAXIS: Patients receive tacrolimus* IV once daily (QD) or orally (PO) BID on days 5-180. Patients also receive mycophenolate mofetil PO thrice daily (TID) or IV on days 5-35. Treatment with tacrolimus and mycophenolate mofetil may continue in the presence of active GVHD.

*NOTE: Patients intolerant of tacrolimus may receive cyclosporine.

After completion of study treatment, patients are followed up twice weekly for 100 days, twice monthly until 6 months, monthly until the patient is off immunosuppressive therapy without evidence of GVHD, and then at least yearly for a total of 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Eligible patients will have a histopathologically confirmed diagnosis of hematologic malignancy in one of the following categories:

  * Acute myelogenous leukemia

    * In first complete remission (CR1) with poor risk cytogenetics according to National Comprehensive Cancer Network (NCCN) guidelines for acute myeloid leukemia (AML): monosomal karyotype, -5, 5q-,-7,7q-, inv (3), t(3;3), t(6;9), t(9;22) and complex karyotypes (>= 3 unrelated abnormalities [abn]) and normal cytogenetics with fms-related tyrosine kinase 3 (FLT3)-internal tandem duplications (ITD) mutation
    * In pediatrics, all of the above and 11q23-non t(9;11)
    * In second complete remission (CR2) or third complete remission (CR3)
    * With chemosensitive primary refractory disease
  * Acute lymphocytic leukemia

    * In CR1 with poor risk cytogenetics:

      * For adults according to NCCN guidelines for acute lymphoblastic leukemia (ALL): hypoploidy (< 44 chromosomes); t(v;11q23): mixed lineage leukemia (MLL) rearranged; t(9;22) (q34;q11.2); complex cytogenetics (5 or more chromosomal abnormalities); high white blood cell (WBC) at diagnosis (>= 30,000 for B lineage or >= 50,000 for T lineage)
      * For pediatrics t(9;22), intrachromosomal amplification of chromosome 21 (iAMP21)loss of 13q, and abnormal 17p
    * In CR2 or CR3
    * With chemosensitive primary refractory disease
  * Myelodysplastic syndrome in high-intermediate (int-2) and high risk categories
* Karnofsky or Lansky performance status >= 80
* A pretreatment measured creatinine clearance (absolute value) of >= 50 ml/minute
* Serum bilirubin =< 2.0 mg/dl
* Serum glutamic oxaloacetic transaminase (SGOT) and serum glutamate pyruvate transaminase (SGPT) =< 2.5 times the institutional upper limits of normal
* Ejection fraction measured by echocardiogram or multigated acquisition scan (MUGA) >= 50%
* Diffusing capacity of the lung for carbon monoxide (DLCO) and forced expiratory volume in one second (FEV1) > 60% predicted
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control or abstinence) prior to study entry and for six months following duration of study participation; should a woman become pregnant or suspect that she is pregnant while participating on the trial, she should inform her treating physician immediately
* The recipient must have a related donor genotypically human leukocyte antigen (HLA)-A, B,C and DRB1 loci haploidentical to the recipient
* No HLA matched sibling or matched unrelated donor is available
* Patients should be off all previous intensive therapy, chemotherapy or radiotherapy for 3 weeks prior to commencing therapy on this study

  * (NOTE: Low dose chemotherapy or maintenance chemotherapy given within 7 days of planned study enrollment is permitted; these include: hydroxyurea, 6-meraptopurine, oral methotrexate, vincristine, oral etoposide, and tyrosine kinase inhibitors [TKIs]; FLT-3 inhibitors such as sorafenib, crenolanib, quizartinib, midostaurin can also be given up to 3 days before conditioning regimen)
* Adequate organ function
* All subjects must have the ability to understand and the willingness to sign a written informed consent
* Prior radiation therapy that would exclude the use of TMLI

DONOR ELIGIBILITY CRITERIA:

* DONOR: Age =< 60 years of age
* DONOR: For younger donors, no more than 20 mL bone marrow may be harvested per kg of donor body weight
* DONOR: Medical history and physical examination confirm good health status as defined by institutional standards
* DONOR: Seronegative for human immunodeficiency virus (HIV) antigen (Ag), HIV 1+2 antibody (Ab), human T-lymphotropic virus (HTLV) I/II Ab, hepatitis B surface antigen (HBsAg), hepatitis B core antibody (HBcAb) (immunoglobulin [Ig]M and IgG), hepatitis C virus (HCV) Ab, rapid plasma reagin (RPR) for syphilis within 30 days of apheresis collection
* DONOR: Genotypically haploidentical as determined by HLA typing, preferably a non-maternal HLA haploidentical relative; eligible donors include biological parents, siblings or half siblings, or children
* DONOR: Female donors of child-bearing potential must have a negative serum or urine beta-human chorionic gonadotropin (HCG) test within three weeks of mobilization
* DONOR: The donor must have been informed of the investigational nature of this study and have signed a consent form in accordance with federal guidelines and the guidelines of the participating institution
* DONOR: Selection of a haploidentical donor will require absence of pre-existing donor-directed anti-HLA antibodies in the recipient

Exclusion Criteria:

* Patients should not have any uncontrolled illness including ongoing or active bacterial, viral or fungal infection
* Patients may not be receiving any other investigational agents, or concurrent biological, intensive chemotherapy, or radiation therapy for the previous three weeks from conditioning

  * (NOTE: Low dose chemotherapy or maintenance chemotherapy given within 7 days of planned study enrollment is permitted; these include: hydroxyurea, 6-meraptopurine, oral methotrexate, vincristine, oral etoposide, and tyrosine kinase inhibitors [TKIs]; FLT-3 inhibitors such as sorafenib, crenolanib, quizartinib, midostaurin can also be given up to 3 days before conditioning regimen)
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to any in the pre- or post-transplant regimen
* Pregnant women are excluded from this study
* Patients with other active malignancies are ineligible for this study, other than non-melanoma skin cancers
* The recipient has a medical problem or neurologic/psychiatric dysfunction which would impair his/her ability to be compliant with the medical regimen and to tolerate transplantation or would prolong hematologic recovery which in the opinion of the principal investigator would place the recipient at unacceptable risk
* Patients may not have had a prior autologous or allogeneic transplant
* HLA-matched or partially matched (7/8 or 8/8) related or unrelated donor is available to donate
* Patients may not have received more than 3 prior regimens, where the regimen intent was to induce remission
* Patients treatment history may not include anti-CD33 monoclonal antibody therapy (e.g., SGN-CD33 or Mylotarg)
* Subjects, who in the opinion of the investigator, may not be able to comply with the safety monitoring requirements of the study

DONOR EXCLUSION CRITERIA:

* DONOR: Evidence of active infection
* DONOR: Medical or physical reason which makes the donor unlikely to tolerate or cooperate with growth factor therapy and leukapheresis
* DONOR: Factors which place the donor at increased risk for complications from leukapheresis or granulocyte-colony stimulating factor (G-CSF) therapy
* DONOR: HIV positive

Ages: 12 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 31 (Actual)
Dates: Start 2015-06-25 (Actual); Primary Completion 2025-05-20 (Actual); Study Completion 2025-05-20 (Actual)

PRIMARY OUTCOMES:
Incidence of dose-limiting toxicity (DLT) scored on both the Bearman Scale and National Cancer Institute Common Terminology Criteria for Adverse Events version 4.03 | Up to 100 days
  Toxicity information recorded will include the type, severity, and the probable association with the study regimen. Tables will be constructed to summarize the observed incidence by severity and type of toxicity.
Maximum tolerated dose of TMLI when given in combination with fludarabine phosphate and cyclophosphamide, defined as the highest dose where 6 patients have been treated and at most one patient experiences DLT | Up to day -3
  Toxicity information recorded will include the type, severity, and the probable association with the study regimen. Tables will be constructed to summarize the observed incidence by severity and type of toxicity.

SECONDARY OUTCOMES:
Complete remission proportion | At day 30
Immune reconstitution of B, T and NK cells | Up to 1 year
Incidence of acute GVHD of grades 2-4 and 3-4 | Within the first 100 days post-transplant
  The cumulative incidence of relapse/progression, non-relapse mortality and acute/chronic GVHD will be calculated as competing risks.
Incidence of chronic GVHD | After 180 days post-transplant assessed up to 5 years
  The cumulative incidence of relapse/progression, non-relapse mortality and acute/chronic GVHD will be calculated as competing risks.
Incidence of infection | Up to day 100
  Microbiologically documented infections will be reported by site of disease, date of onset, severity and resolution, if any.
Minimal residual disease | Up to 180 days post-transplant
Non-relapse mortality (NRM) | Up to 5 years
  The cumulative incidence of relapse/progression, non-relapse mortality and acute/chronic GVHD will be calculated as competing risks.
Overall survival | Time from start of protocol therapy to death, or last follow-up, whichever comes first, assessed up to 5 years
  Survival estimates will be calculated using the Kaplan-Meier method.
Progression-free survival | Time from start of protocol therapy to death, relapse/progression, or last follow-up, whichever comes first, assessed up to 5 years
  Survival estimates will be calculated using the Kaplan-Meier method.
Incidence of grade 3-5 adverse events per CTCAE v4.03 | Up to 100 days post-transplant
  Toxicity information recorded will include the type, severity, and the probable association with the study regimen. Tables will be constructed to summarize the observed incidence by severity and type of toxicity.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Rosenthal, Principal Investigator — City of Hope Comprehensive Cancer Center
Locations (1):
- City of Hope Comprehensive Cancer Center, Duarte, California, United States